CLINICAL TRIAL: NCT03985319
Title: A Randomized, Open-label, Cross-over Design Clinical Trial to Assess the Pharmacokinetic/Pharmacodynamic Properties and Safety of YYD601 20mg After Oral Administration in Healthy Adult Subjects (Phase1)
Brief Title: Clinical Trial to Assess the PK/PD of YYD601 20mg After Oral Administration if Healthy Adult Subjects (Phase1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YYPCT_YYD601_P1(2)
Record Dates: First submitted 2019-05-29; First posted 2019-06-13 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Drugs, Investigational; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YYD601 20mg (Experimental): Esomeprazole IR 10mg + esomeprazole SR 10mg
  Interventions: Drug: Nexium tab 20mg
- Nexium tab 20mg (Active Comparator): Esomeprazole magnesium trihydrate 22.3mg. Astrazeneca
  Interventions: Drug: YYD601 20mg

INTERVENTIONS:
Drug: YYD601 20mg — Esomeprazole IR 10mg + Esomeprazole SR 10mg (Expected efficacy and effects: GERD)
  Other Names: Experimental drug
  Arms: Nexium tab 20mg
Drug: Nexium tab 20mg — Esomeprazole magnesium trihydrate 22.3mg Effecacy and Effects: GERD and Antibiotics combined therapy to eradicate the Helicobacter pylori
  Other Names: comparator drug
  Arms: YYD601 20mg

SUMMARY:
Clinical Trial to Assess the PK/PD of YYD601 20mg After Oral Administration if Healthy Adult Subjects (Phase1)

DETAILED DESCRIPTION:
To evaluate comparatively a characteristics and safety of the PK/PD of single/repeated oral administration YYD601 20mg and Nexium tab 20mg and the effects of food influence the PK/PD of YYD601 20mg in a healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of over 19 years old at the time of screening.
* Volunteers weighing over 50 kg with ideal body weight (IBW) between -20% ~ 20%
* Subjects don't have congenital or chronic disease and is without pathologic symptom or finding on medical exam.
* Subjects evaluated eligible for the study based on the screening test results such as laboratory tests including serology, hematology, blood chemistry and urinalysis, etc and electrocardiogram(ECG).
* Subejctys who signed on the written informed consent form and comply with study requirements after listening adn fully understanding the details of this study.

Exclusion Criteria:

* Who has hyper sensitivity reaction about other drugs, ingredients, components of investigator product or compound of benzimidazole.
* Who has genetic problem like fructose tolerance, glucose-galctose absorption, deficiency or sucrase-iso maltase deficiency.
* Medical history or evidence (hepatobiliary, renal, cardiovascular, endocrine, respiratory, gastrointestinal, hemato-oncology, central nervous system, psychiatric and musculoskeletal system) that can affect absorption, distribution, metabolism and excretion of a given drug.
* Subject who has over 141mmHg or under 89mmHg of systolic pressure or over 95mmHg of diastolic pressure in vital sign or over 100 times/min of pulse rate.
* Who has active liver disease, (AST, ALT, total bilirubin > 2 x LNR), (BUN, creatinine >1.5 x LNR) or clinically abnoramal result at screening test.
* Creatinine clearance < 80 mL/min (calcaulated by Cockcroft-Gault formula using serum creatinine)
* History of gastrointestinal disease (e.g., Crohns disease, active peptic ulcer) or gastrointestinal surgery that may affect the absorption of the study drug (excluding simple appendectomy or herniorrhaphy)
* Treatments for peptic ulcer, esophageal disease, Zollinger-Ellison syndrome diagnosis therapy or clinically related histories within 3 months prior to the first dose.
* Positive 13C-urea breath test
* A history of serious trauma within 4 weeks, or resection operation (exculding simiple appendectomy or herniorrhaphy) and/or relevant history or laboratory or clinical findings indicative of acute disease.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Cmax | Integrated gastric acidity: Stomach acid test (24pH) on 1 day, 5 day, 11 day, 16 day
  Cmax after single administration and repeated administration
AUC | Integrated gastric acidity: Stomach acid test (24pH) on 1 day, 5 day, 11 day, 16 day
  AUC after single administration and repeated administration

SECONDARY OUTCOMES:
AUC | pH>4(%): stomach acid test(24pH) on -1 day, 5 day, 11 day, 16 day and change in serum gastrin level on -1 day, 1day, 5 day
  AUC after single administration and repeated administration
Tmax | pH>4(%): stomach acid test(24pH) on -1 day, 5 day, 11 day, 16 day and change in serum gastrin level on -1 day, 1day, 5 day
  Tmax after single administration and repeated administration
t1/2 | pH>4(%): stomach acid test(24pH) on -1 day, 5 day, 11 day, 16 day and change in serum gastrin level on -1 day, 1day, 5 day
  t1/2 after single administration and repeated administration

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook national university hospital, Daegu, South Korea

REFERENCES:
- [Derived] Lee HW, Kang WY, Park JS, Lee JH, Park JJ, Gwon MR, Yoon YR, Seong SJ. A Pharmacokinetic/Pharmacodynamic Study of Esomeprazole Comparing a Dual Delayed-Release Formulation (YYD601) to a Conventional Formulation Following Multiple Administrations in Healthy Adult Subjects. Drug Des Devel Ther. 2025 Jan 8;19:97-110. doi: 10.2147/DDDT.S500253. eCollection 2025. PMID 39803609